CLINICAL TRIAL: NCT00018317
Title: Resistance Training and Diet in Patients With Chronic Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: AGCG-005-99F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Kidney Failure, Chronic
Keywords: Diet; exercise
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Diet, Protein-Restricted; Resistance Training; Exercise

INTERVENTIONS:
Behavioral: low protein diet
Behavioral: resistance training
Behavioral: combination of diet control and exercise

SUMMARY:
This study will examine the effects of long-term adherence to a low protein diet (LPD) of 0.6 g/kg-1/d-1 with and without progressive resistance exercise training in patients with impaired renal function on body composition, renal function (glomerular filtration rate), nitrogen balance, muscle strength and size, and functional capacity. The hypothesis is that adherence to a LPD will result in a reduction in skeletal muscle mass and reduced strength and functional capacity while those patients who adhere to the LPD and exercise will demonstrate a similar preservation of renal function but will have greater fat free mass, muscle mass and strength. The intervention trial will last 18 months in which patients with moderate renal failure will be randomly assigned to one of 4 interventions: standard care, standard care + exercise, LPD, and LPD with exercise. In this way the independent and combined effects of diet and exercise on the progression of renal disease and body composition will be monitored. This study will have important implications for the treatment of patients with chronic renal failure. New strategies of combining exercise with recommendations of a low protein diet may slow the progression of renal disease and improve strength and functional capacity in these at-risk patients.

DETAILED DESCRIPTION:
Management of dietary protein intake of the CRF patient represents a critical balance between providing adequate protein to meet nutritional requirements, and limiting protein intake in the hope of slowing or abating the progression of CRF. A number of studies have demonstrated that reduced dietary protein intake can slow the progression of chronic renal failure. Finding effective ways to increase nitrogen retention and decrease urinary nitrogen excretion may help CRF patients maintain a more positive nitrogen balance and lessen the nitrogen load on the kidneys for a given dietary protein intake. Our laboratory has demonstrated that in older men and women, the consequence of adherence to a low protein diet is an accommodation that results in decreased muscle mass, strength,and compromised immune function. We have also demonstrated that when healthy, free living older men and women consume a weight maintenance diet providing the RDA for protein of 0.8 g/kg-1/day-1 for 15 weeks they lose skeletal muscle mass. These data clearly indicate that elderly people have an increased need for dietary protein (compared to young people). Data has also demonstrated that progressive resistance exercise improves nitrogen balance in older healthy individuals as well as in patients with mild to moderate chronic renal failure.

ELIGIBILITY:
* Men and women 50-89 years with chronic renal failure (defined as creatinine clearance of 25-65).
* Volunteers must be able to fulfill the requirements associated with this protocol.
* Volunteers may be hypertensive and/or diabetic.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Chatoth, M.D.
Locations (1):
- Central Arkansas Veterans Healthcare System, Little Rock, Arkansas, United States